CLINICAL TRIAL: NCT06520930
Title: The Effect of the Structured Supportive Approach Based on Kolcaba Comfort Theory Applied to Primiparous Pregnant Women on the Comfort Level in the Last Trimester
Brief Title: The Effect of Breathing Exercises on Comfort Level in Primiparous Pregnant Women
Acronym: breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Kucuk (Other)
Responsible Party: Sponsor-Investigator, Sibel Kucuk, lecturer, Harran University
Organization: Harran University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HRN-SK-44
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Primipara Pregnant
Keywords: primipara pregnant; comfort; breathing therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment two groups
Who Masked: Participant
Masking Description: statistical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms (No Intervention): First Stage: As a pre-test, pulse, respiratory rate and saturation values will be checked, Descriptive Questionnaire and General Comfort Scale (GAS) will be applied to primiparous pregnant women in the control group.
  Second Stage: As the final test, the heart rate, respiratory rate, blood pressure and saturation values will be checked again at the end of the 8th session for primiparous pregnant women, and the Descriptive Questionnaire and General Comfort Scale (GAS) will be applied.
- Intervention Group (Experimental): As a pre-test, pulse, respiratory rate, blood pressure and saturation values will be checked, Descriptive Questionnaire and General Comfort Scale (GAS) will be applied to the primiparous pregnant women in the experimental groups. Breathing therapy exercises based on Kolcaba's comfort theory were designed as face-to-face training by the researcher himself, who received breathing therapy training for primiparous pregnant women once a week, for a total of 8 sessions. 6 pieces will be created within the session. Each session lasts approximately 45-60 minutes. As the final test, pulse, respiratory rates, blood pressure and saturation values will be checked again at the end of the 8th session/week to determine the change in primiparous pregnant women, and the Descriptive Questionnaire and General Comfort Scale (GAS) will be applied.
  Interventions: Behavioral: breathing exercise therapy

INTERVENTIONS:
Behavioral: breathing exercise therapy — Description: The breathing exercises to be applied were taught to each pregnant woman face to face with one-on-one training. The taught practice was then repeated by the pregnant woman and the researcher together. In the next step, pregnant women were asked to perform the application themselves. In this way, it was determined whether individual breathing exercise practices were performed correctly and effectively. After the one-on-one training was completed, the pregnant women were divided into groups of maximum six people and breathing exercise exercises were performed 7 days a week, once a day and once a week face-to-face for 8 weeks. Each session lasted approximately 45 minutes. For 8 weeks, a short reminder message was sent to pregnant women every morning to ensure that they did not interrupt their daily breathing exercise practices, and they were called in the evening to check whether they had performed the application correctly and whether they had any problems.
  Arms: Intervention Group

SUMMARY:
Pregnancy is a special period in which some changes occur in bio-psycho-social areas and adaptation to these changes is achieved (Üzar and Erkan; 2019). While this special period creates happiness and peace in some women, it can cause emotional and relational changes in some women, create anxiety and anxiety, and negatively affect their comfort level (Al-Mutawtah et al., 2023; Yar and Yılmaz, 2021). In order to reduce the effects of complaints experienced during pregnancy and ensure adaptation, nurses who provide holistic, innovative, effective and supportive care, determine the comfort needs of the individual and the family, and improve their comfort levels by planning and applying interventions specific to the areas needed.

It increases. (Arslankılıç and Göl, 2020; Kolcaba1991). In this context, breathing exercises, which are defined as an invisible spirit that provides the connection between body, mind and soul, gives life to its owner, has an important place in order to increase the comfort level and ensure adaptation to the pregnancy process (Kartal, 2018). Because breathing exercises stimulate the parasympathetic nervous system, increase blood oxygenation and, as a result, trigger the secretion of endorphins. The increased release of endorphins reduces the heart rate, resulting in a feeling of calm. In addition, endorphin suppresses the sympathetic nervous system and reduces the release of cortisol, the stress hormone, thus keeping psychotic emotions under control (Issac, et al., 2023).Thus, the complaints that occur during pregnancy can be minimized with correct and effective breathing techniques and the comfort level can be increased. As a result of literature reviews; Regular breathing exercises increase lung volume, increase the endurance and efficiency of the diaphragm muscle, reduce dyspnea, provide easier breathing, and help eliminate bronchial secretions (Özulus, 2018; Tucker and Jenkins 1996). It has been found that it is effective in reducing hypertension, fatigue and anxiety, and that a 30-session intervention lasting 5 minutes per day for women who have given birth prematurely significantly reduces anxiety (Ölçer and Oskay; 2015; Chang et al., 2009). For this reason, the concept of comfort should be evaluated multidimensionally during pregnancy and holistic nursing interventions should be implemented to increase the comfort level.

In this study, it is envisaged that breathing exercise practices will increase the general comfort level of primiparous women, such as adaptation to pregnancy, increase in sleep quality, decrease in pain, decrease in anxiety levels, improvement in vital signs and conscious management of third trimester changes. At the same time, these research findings will constitute an important data source in research on the general comfort level effectiveness of breathing exercises to be performed on primiparous pregnant women from the 2nd trimester onwards in the 3rd trimester. Because, no randomized controlled study has been conducted in Turkey regarding the effect of breathing exercise on the general comfort level of last trimester pregnant women.

DETAILED DESCRIPTION:
The population of the research consists of primiparous women who applied to the Private Metrolife Hospital Obstetrics and Gynecology outpatient clinic. The sample size of the study was determined using post hoc power analysis G-Power 3.1.9.4 program. In the power analysis conducted for the research, it was determined that a total of 72 primiparous women, including at least 36 people in both groups, were included in the study in order to reach a 95% confidence interval, an effect size of 0.6, an α-type error estimate of 0.05 and 80% power in the experimental and control groups with the pretest-posttest. It was determined that there was a need for inclusion. In view of the possibility that primiparous pregnant women who will participate in the study may withdraw from the study for various reasons, the total number of primiparous pregnant women was determined as 80, 40 for the control group and 40 for the experimental group. The research was completed with 40 primiparous pregnant women in the intervention group and 40 primiparous pregnant women in the control group, according to the CONSORT flow chart.

The breathing exercises to be applied were taught face to face to each pregnant woman by the researcher who has a "Breathing Therapy" certificate. The taught practice was then repeated by the pregnant woman and the researcher together. In the next step, pregnant women were asked to perform the application themselves. In this way, it was determined whether individual breathing exercise practices were performed correctly and effectively. After the one-on-one training was completed, the pregnant women were divided into groups of maximum six people and breathing exercise exercises were performed 7 days a week, once a day and once a week face-to-face for 8 weeks. Breathing exercises were administered face to face to a maximum of two groups per day, and each session lasted approximately 45 minutes. In addition, for 8 weeks, a short reminder message was sent to pregnant women every morning (between 10:00-11:00) to prevent them from disrupting their daily breathing exercise practices, and they were called in the evening (between 17:00-18:00) to check whether they had performed the application correctly or not. It was checked whether they were experiencing any problems.

Data collection tools; Introductory Information Form: This form was prepared by the researcher by scanning the relevant literature; Socio-demographic characteristics of primiparous pregnant women (age, age at marriage, duration of marriage, education level, profession, income level, social security status, place of residence, family structure), obstetric characteristics (gestational age, planned pregnancy, problems experienced during pregnancy, any relaxing practice) and pulse, respiratory rate and saturation values were checked.

General Comfort Scale (GAS) was used. The intervention group had data collection tools filled out before and after therapy.

Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Volunteer to participate in the study, Those aged 19 and over, non-smoker Without a risky pregnancy diagnosis (without obstetric complications, psychiatric diagnosis, ear, nose or throat problems and systemic disease) Literate and without communication difficulties 2nd trimester primiparous pregnant women who are 21st week of pregnancy and later

Exclusion Criteria:

They want to withdraw from the research at any point during the research. Those who accept face-to-face application and then give up or do not continue the application, Not doing daily breathing exercises, Couldn't be reached by the researcher even though he called at most three times a day, Changing hospital, Women who fill out the research data collection forms incompletely will be excluded from the sample.

-

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — primiparous pregnant women
Enrollment: 80 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | Pregnant women in the experimental and control groups will be evaluated with the start of the study
  socio-demographic characteristics of primiparous pregnant women (age, age at marriage, duration of marriage, education level, profession, income level, social security status, place of residence, family structure), obstetric characteristics (gestational age, planned pregnancy, pregnancy It will be used to obtain information about the problems experienced, any relaxing practice during pregnancy) and pulse, respiratory rate and saturation values.

SECONDARY OUTCOMES:
General Comfort Scale (GAS) | It will be filled out before starting the study for the experimental and control groups, and will be filled in again to compare both groups in the 3rd trimester after the training is completed for the experimental group in the 8th week.
  The general comfort scale was developed by Katherine Kolcaba in 1992. The Turkish validity and reliability study of the scale was conducted by Kuğuoğlu and Karabacak (2008). The scale is a four-point Likert type and consists of a total of 48 items. Comfort levels of the scale; relief (16 items), relaxation (17 items) and overcoming problems (15 items). The response patterns of the scale, which consists of positive and negative items, are given in a mixed manner. Accordingly, in positive items, a high score (4) indicates high comfort and a low score (1) indicates low comfort. In the evaluation of the scale, the negative scores obtained (5, 6, 8, 12, 13, 14, 18, 19, 20, 21, 22, 24, 2526, 28, 32, 34, 35, 39, 40, 41, 42, 45, 48) are reverse coded and summed with positive items. The highest total score that can be obtained from the scale is 192, and the lowest total score is 48. Low comfort is expressed with one point, high comfort with four points. In the validity and reliability study, t

CONTACTS AND LOCATIONS:
Overall Officials: SİBEL KÜÇÜK, Lecturer, Principal Investigator — Harran University
Locations (1):
- Harran University, Sanliurfa, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Mutawtah M, Campbell E, Kubis HP, Erjavec M. Women's experiences of social support during pregnancy: a qualitative systematic review. BMC Pregnancy Childbirth. 2023 Nov 10;23(1):782. doi: 10.1186/s12884-023-06089-0. PMID 37950165